CLINICAL TRIAL: NCT00967343
Title: An Open-label, Uncontrolled, Multicenter, Multinational Study on the Efficacy and Safety of Administration of Donor Lymphocytes Depleted of Alloreactive T-cells (ATIR), Through the Use of TH9402 and Light Treatment in an ex Vivo Process, in Patients Receiving a CD34-selected Peripheral Blood Stem Cell Graft From a Related, Haploidentical Donor
Brief Title: Efficacy and Safety of a Donor Lymphocyte Preparation Depleted of Functional Host Alloreactive T-cells (ATIR) in Patients Undergoing a Peripheral Blood Stem Cell Transplant From a Related, Haploidentical Donor
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR-AIR-004; EudraCT no. 2008-008198-73
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Myeloid Leukemia; Lymphoblastic Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome; Myeloproliferative Disorders
Keywords: Haploidentical stem cell transplantation; Graft-versus-host disease; Immune reconstitution; Alloreactive T-cells; Photodepletion; TH9402; Transplant related mortality; Hematologic malignancy
MeSH Terms: conditions — Leukemia, Myeloid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATIR (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of host functional alloreactive T-cells

INTERVENTIONS:
Biological: Donor lymphocyte preparation depleted of host functional alloreactive T-cells — Single intravenous infusion with 2x10E6 T-cells/kg

SUMMARY:
The purpose of this study is to determine whether the administration of a donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR) after a T-cell depleted stem cell transplant from a related, haploidentical donor enhances survival by improving the immune effect against infections while preventing graft-versus-host disease .

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation is the treatment of choice for many patients with leukemia and other hematologic malignancies. However, a major limitation of this therapy is that for a significant number of patients no fully HLA-matched donor can be found. The application of partially HLA-matched (haploidentical) family donors, who are virtually always available, has some complications. If there is no T-cell add-back it increases the risk for life-threatening infections and disease relapse, while in case of T-cell add-back the risk for graft-versus-host disease is raised.

Kiadis Pharma has developed a method to selectively deplete host alloreactive T-cells through photodynamic therapy, using TH9402 ex vivo. The donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR) is administered to the patient 28-42 days after the stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

One of the following hematological malignancies:

* Acute Myeloid Leukemia (AML)
* Acute Lymphoblastic Leukemia (ALL)
* Myelodysplastic Syndrome (MDS)
* Ph-positive chronic myeloid leukemia (CML)
* Non-Hodgkin Lymphoma (NHL)
* Myelodysplastic Syndrome (MDS)
* Chronic Myeloid Leukemia (CML)
* Multiple Myeloma (MM)
* Chronic Lymphocytic Leukemia (CLL)
* Myeloproliferative Syndrome (MPS)

Exclusion Criteria:

* AML in 1st complete remission with good risk karyotypes
* MM featuring concurrent extramedullar disease or being non-responsive to prior therapy
* CML in blast crisis
* CLL concurrently transformed into high-grade lymphoma and failing to demonstrate at least partial remission
* NHL with concurrent bulky disease (≥ 5 cm)
* Diffusing Capacity for Carbon Monoxide (DLCO) < 40% predicted
* Left ventricular ejection fraction < 40%
* AST/SGOT > 2.5 x ULN
* Bilirubin > 1.5 x ULN
* Creatinine > 1.5 x ULN
* HIV positive
* Positive pregnancy test for women of childbearing age
* Prior haploidentical peripheral blood stem cell or cord blood transplantation
* Less than 2 years from a prior allogeneic stem cell transplantation
* Estimated probability of surviving less than three months
* Major anticipated illness or organ failure incompatible with survival from transplant
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and informed consent impossible
* Known allergy to any of the components of ATIR
* Any other condition which, in the opinion of the investigator, makes the patient ineligible for the study

Donor Inclusion Criteria:

* Haploidentical family donor with 2 to 3 mismatches at the HLA-A, -B and/or DR loci of the unshared haplotype.
* Male or female, age ≥ 16, ≤ 75 years.
* Donors must be fit to receive G-CSF and undergo apheresis (normal blood count, normotensive and no history of stroke).
* Donor must have Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
* Donor must provide written informed consent.

Donor Exclusion Criteria:

* Medically uncontrolled coronary heart disease.
* Myocardial infarction within the last 3 months.
* History of uncontrolled seizures.
* History of malignancy (except basal cell or squamous carcinoma of the skin, positive PAP smear and subsequent negative follow up).
* Positive test result for any of the mandatory viral tests in the applicable region, except for a positive cytomegalovirus (CMV) result, which does not lead to exclusion.
* Presence of a transmissible disease (such as HIV positive), a major illness, a suspected systemic dysfunction and/or an active inflammatory or autoimmune disorder.
* Female donors who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Mielke, MD, Study Chair — Julius Maximilian University of Würzburg, Germany; Denis-Claude Roy, MD, Study Chair — Maisonneuve-Rosemont Hospital, Montreal, Canada; Andrea Velardi, MD, Principal Investigator — University Of Perugia; Katy Rezvani, MD PhD, Principal Investigator — Hammersmith Hospital, London, United Kingdom
Locations (15):
- Ohio State University, Comprehesive Cancer Center, Columbus, Ohio, United States
- Belgium (4):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Université Libre de Bruxelles - Institute Jules Bordet, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - University of Liege - CHU Sart Tilman, Liège
- Canada (3):
  - HHSC, Henderson Hospital Site, Hamilton, Ontario
  - Ontario Cancer Institute / Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- Germany (4):
  - Universitätsklinikum Freiburg, Medizinische UNI-Klinik, Freiburg im Breisgau
  - Universitätsklinikums Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Mainz, Mainz
  - Universitätsklinikum Würzburg, Würzburg
- Perugia University, Perugia, Italy
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATIR
Started | 40
Completed | 2
Not Completed | 38
Not completed — Study termination by sponsor | 12
Not completed — Death | 24
Not completed — Relapse | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATIR
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Hematologic malignancy [Count of Participants; unit: Participants]
  Acute lymphatic leukemia | 5
  Acute myeloid leukemia | 22
  Chronic myeloid leukemia | 1
  Myelodysplastic syndrome | 3
  Myeloproliferative syndrome | 1
  Other acute leukemia | 2
  Other leukemia | 3
  Plasma cell disorder | 3
Donor HLA compatibility (HLA-A, -B, -DR) [Count of Participants; unit: Participants]
  Donor HLA compatibility (HLA-A, -B, -DR): 3/6 | 27
  Donor HLA compatibility (HLA-A, -B, -DR): 4/6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Transplant Related Mortality
Description: TRM is defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. accident, suicide)
Time Frame: 6, 12 and 24 months after the transplantation
Measure: Number; unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 40
Kaplan-Meier estimates (%)
  TRM at 6 months post HSCT | 33
  TRM at 12 months post HSCT | 56
  TRM at 24 months post HSCT | 71

2. Secondary Outcome: Incidence and Severity Graft-versus-host Disease (GVHD)
Description: GVHD was graded according to standard criteria as referred to in the reference module (Filipovich et al. 2005; Przepiorka et al. 1995).
Time Frame: Up to 24 months after the transplantation
Measure: Number; unit: Percentage of participants
Arm/Group | ATIR
Number analyzed (Participants) | 40
Percentage of participants
  Grade II acute GVHD (moderate) | 7.5
  Grade III (moderate) or IV (severe) acute GVHD | 12.5
  Severe chronic GVHD | 5

3. Secondary Outcome: Progression Free Survival
Time Frame: Up to 24 months after the transplantation
Population: Data were not collected, premature termination of study
Arm/Group | ATIR
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence and Severity of Bacterial, Viral or Fungal Infection
Time Frame: Up to 24 months after the transplantation
Population: Data not collected, premature termination of study
Arm/Group | ATIR
Number analyzed (Participants) | 0

5. Secondary Outcome: Immune Reconstitution
Time Frame: Up to 24 months after the transplantation
Population: Data were not collected, premature termination of study
Arm/Group | ATIR
Number analyzed (Participants) | 0

6. Secondary Outcome: Health Status (Including Quality of Life)
Time Frame: Up to 24 months after the transplantation
Population: Data were not collected, premature termination of study
Arm/Group | ATIR
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival
Time Frame: 6, 12, and 24 months after the transplantation
Measure: Number; unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 40
Kaplan-Meier estimates (%)
  OS 6 months after the HSCT | 65
  OS 12 months after the HSCT | 33
  OS 24 months after the HSCT | 22

ADVERSE EVENTS:
Arm/Group | ATIR
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR (N=40)
Acute graft versus host disease (Immune system disorders) | 3
Chronic graft versus host disease (Immune system disorders) | 1
Bacterial sepsis (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
JC virus infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hepatitis failure (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR (N=40)
Acute graft versus host disease (Immune system disorders) | 4
Cytomegalovirus infection (Infections and infestations) | 2
abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No